CLINICAL TRIAL: NCT05707117
Title: Effects of Tendon Neuroplastic Training (TNT) on Pain and Strength in Lateral Epicondylitis.
Brief Title: Effects of Tendon Neuroplastic Training (TNT) in Lateral Epicondylitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah IU Muhammad Hamza khan
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Tendon neuroplastic training; strength training
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Tendon neuroplastic training (TNT) (Experimental): the strength training of the wrist extensors are being done with the help of an externally pace device
  Interventions: Other: Tendon neuroplastic training (TNT)
- Group B: Conventional treatment (Active Comparator): static stretching and myofascial release on wrist extensors
  Interventions: Other: group B Conventional treatment

INTERVENTIONS:
Other: Tendon neuroplastic training (TNT) — Subjects will attend physical therapy for three non-consecutive days per week for a total 4 consecutive weeks. Exercise would involve isolated flexion, extension with a dumbbell. This exercise would be paced with external audio/visual cue on smart phone using proMetronome app. Patients will listen to the sound and track the movement of metronome with the eyes. Pace of metronome will be set at 20 beats per minute such that each beat will be 3 sec apart. This will allow a 3sec concentric and 3 sec eccentric phases.4 sets of 8 repetitions would be completed with a 2-minute rest between each set. Exercise will begin with 3 pounds weight, but it would be made sure that this wouldn't cause pain during exercise (more than 5/10), gradual progression in weight to 5 pounds after 2nd weeks.
  Arms: Group A: Tendon neuroplastic training (TNT)
Other: group B Conventional treatment — Subjects assigned to this group will undergo static stretching of Extensor carpi radialis brevis and myofascial release for 4 weeks, 3 sessions a week. Myofascial release technique will be applied for 5 minutes and 2 reptations per session
  Arms: Group B: Conventional treatment

SUMMARY:
The aim of this research is to determine effects tendon neuroplastic training on strength, pain, and function in lateral epicondylitis. Randomized controlled trials will be conduct in National Institute of Rehabilitation Medicine Islamabad and Lady Reading Hospital Peshawar. The sample size is 34. The subjects will be divided in two groups, 17 subjects in tendon neuroplastic training group and 17 subjects will be assigned to conventional exercises group. Study duration is of one year. Sampling technique applied will be non-probability convenient sampling technique. Only 20-45 years old patients diagnosed with lateral epicondylitis will be included. Tools used in the study are Numeric pain scale, Dynamometer for grip strength and Patient rated tennis elbow evaluation for functional status.

DETAILED DESCRIPTION:
Lateral epicondylitis or tennis elbow is the common musculoskeletal degenerative disorder of the extensor origin at the lateral humeral epicondyle. It is the most common overuse syndrome seen in the primary care with the annual incidence of 1% to 3% in general population. This condition is most prevalent in age group of 45-54 years. The condition effect men and women equally. It mostly effects individuals with the history of repetitive wrist extension activities. Lateral epicondylitis is the chronic symptomatic degeneration (tendinosis) of the tendon of extensor muscles of forearm. According to cyriax most common effected muscle in lateral epicondylitis is extensor carpi radialis brevis (ECRB). Patients with lateral epicondylitis present to clinic with chief complaints of decrease grip strength and increase pain which may have a significant effect on their daily life activities.

Conventional treatment primarily focuses on pain management by anti-inflammatory medicine, Ultrasound, phonophoresis, ionophoresis and corticosteroid injection. In literature other physiotherapy approaches documented which includes manual therapy, stretching and strengthening exercises, electrotherapy, taping, shock-wave therapy, and acupuncture. There is greater evidence in favor of strengthening exercises in patients who have symptoms for more than 6 months. Other approaches also focus on eccentric exercises combined with static stretching exercises in treatment of tendinopathies. Isometric exercises are used to manage and reduce tendon pain. But all these interventions merely focus on the peripheral tissue and not address neuromuscular and complex corticospinal adaptation associated with the persistent pain and therefore lead to chronicity and less desirable outcomes. Tendon neuroplastic training (TNT) is proposed to address the central nervous system component and motor deficit of tendinopathies. It combines isometric or isotonic strengthening training with externally paced audio or visual cue provided by metronome rather than self-paced exercise and strongly focus on neuromuscular control with the aim to induce neuroplasticity. Corticospinal excitability and short interval cortical inhibition are factors through which we can measure motor control and is found altered in tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age between 20-45 years
* Pain and Tenderness over the lateral epicondyle
* At least 2 of cozen's test, Maudsley's test and Mill's test will cause pain at lateral epicondylitis.

Exclusion Criteria:

* Open wounds
* Fracture of elbow Humerus, radius, ulna
* Surgical procedure done around the elbow joint.
* Elbow instability.
* Extensor tendon rupture.
* Symptoms of cervical radiculopathy.
* Radial nerve entrapment.
* Major upper limb surgery.
* Tumor or wound
* Compartment syndrome of anconeus muscle.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Numeric pain Rating scale (NPRS) | 4th week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line

SECONDARY OUTCOMES:
Patient rated tennis elbow evaluation (functional status). | 4th week
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is a specific questionnaire designed for lateral epicondylitis to assess pain and function/ disability. The PRTEE is composed of pain and function subscales, determining pain at rest and during certain activities and assessing difficulty when performing specific and usual activities over the past week on a scale of 10 options, respectively. Scores can be calculated separately for subscales and as a total PRTEE score, with 0 indicating no pain and disability, 100 indicating the worst pain and functional disability score
Dynamometer | 4th week
  The protocol consists of three maximal isometric contractions without pain for 5 s with a rest period of at least 60 s. The patient performs three trials of grip strength using their involved hand while maintaining 90° elbow flexion and neutral forearm position. The patient is asked to squeeze the dynamometer as hard as possible without the sensation of pain. According to a study the mean strength of three measurements was recorded in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- National Institute of Rehabilitation Medicine (NIRM), Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan H, Razzaq A, Afridi A, Sheraz S, Awan WA. Innovative neuroplastic healing: tendon Neuroplastic Training role in pain alleviation and boosting strength in lateral epicondylitis: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Oct 10;26(1):949. doi: 10.1186/s12891-025-08328-1. PMID 41073965